CLINICAL TRIAL: NCT05133752
Title: A Multi-Center, Open-Label, Single-Arm, Phase IV Study to Evaluate the Safety and Clinical Efficacy of Oral Administration With Nemonoxacin in Treating Elderly Patients With Community-Acquired Pneumonia
Brief Title: Oral Nemonoxacin in Treating Elderly Patients With CAP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: TaiGen Biotechnology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-873870-05
Record Dates: First submitted 2021-11-08; First posted 2021-11-24 (Actual); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia | interventions — nemonoxacin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Nemonoxacin (Experimental)
  Interventions: Drug: Nemonoxacin

INTERVENTIONS:
Drug: Nemonoxacin — 500 mg, oral administration, once daily for 7-10 days.

SUMMARY:
This study was to evaluate the safety and efficacy of oral nemonoxacin in treating elderly patients (aged ≥ 65 years) with community-acquired pneumonia (CAP).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 years
* Clinical diagnosis of CAP
* Evidence of inflammatory exudates or infiltrates on chest X-ray

Exclusion Criteria:

* Suspect viral pneumonia, aspiration pneumonia, ventilator-associated pneumonia or hospital-acquired pneumonia
* History of hypersensitivity to quinolone or fluoroquinolone

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-09-11 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 after treatment with oral nemonoxacin once daily for 7-10 days | From Visit 1 (Baseline) till Visit 3 (within 24 hr after last dose)

SECONDARY OUTCOMES:
Number of participants with clinical success in the modified intention-to-treat (mITT) population, intention-to-treat (ITT), and clinically evaluable (CE) populations. | Visit 3 (within 24 hr after last dose)

CONTACTS AND LOCATIONS:
Locations (1):
- Tri-Service General Hospital, Taipei, Taiwan